CLINICAL TRIAL: NCT00132483
Title: ExStroke Pilot Trial: Physical Exercise After Acute Ischaemic Stroke
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Bispebjerg Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: ExStroke Pilot Trial
Record Dates: First submitted 2005-08-19; First posted 2005-08-22 (Estimated); Last update posted 2007-10-22 (Estimated); Status verified 2007-10

CONDITIONS: Stroke
Keywords: Physical activity; cerebral infarct
MeSH Terms: conditions — Stroke; Motor Activity; Cerebral Infarction | interventions — Educational Status

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Intervention arm (Experimental)
  Interventions: Behavioral: Instruction in physical training program
- Control (No Intervention)

INTERVENTIONS:
Behavioral: Instruction in physical training program — Instruction in physical training program.
  Arms: Intervention arm

SUMMARY:
Summary

This study will look at physical exercise after acute ischaemic stroke. It is called the ExStroke Pilot Trial.

Physical activity is associated with a lower risk of first-time stroke. It remains unknown if physical activity also is associated with a lower risk of recurrent stroke. Patients with ischaemic stroke have a 30% to 40% risk of a recurrent stroke during a 5 year follow-up. The risk of acute myocardial infarction (MI) and death from vascular disease is approximately 15% each. The impact of lifestyle factors on risk for these events is insufficiently covered in the international scientific literature.

Purpose:

The purpose of the trial is to examine whether the level of physical activity increases in patients who have had an ischemic stroke, when they are informed about physical activity and instructed in a physical training program. The occurrence of new cerebro- and cardiovascular events in the patients will be registered. The patients are randomised to receive oral and written information by a physician and a physiotherapist about physical exercise; or to a control group with no instruction regarding physical exercise. Both groups will receive the best available therapy with regard to secondary stroke prevention and will be informed about lifestyle factors.

Irrespective of which group the patients are randomised to, all patients will receive the best possible established treatment with regard to prevention of thromboses; blood pressure control; lipid lowering agents, if necessary; and information about diet, tobacco smoking, and vitamin supplements.

Study Design:

The patients will be randomised centrally within 90 days after stroke onset, and they will be re-examined at 3, 6, 9, 12, 18, and 24 months. Inclusion criteria are patients with ischaemic stroke, aged 40 years or older. In the pilot trial a number of 300 included patients is wanted.

DETAILED DESCRIPTION:
Physical exercise after acute ischaemic stroke.

The ExStroke Pilot Trial.

A randomised clinical trial.

Investigation group

Principal investigator:

Gudrun Boysen, Professor, DMSc Department of Neurology Bispebjerg University Hospital

Co-investigators:

2400 Copenhagen NV

Anders Pedersen, Project Nurse

Lars-Henrik Krarup, MD

Thomas Truelsen, MD Ph.D.

Lotte Hansen, Physiotherapist

Marianne Lindahl, Physiotherapist

Christian Gluud, DMSc Copenhagen Trial Unit Rigshospitalet 2100 Copenhagen Ø

Introduction:

Physical activity is associated with a lower risk of first-time stroke. It is unknown if physical exercise reduces risk of recurrent stroke. Clinicians treating stroke patients are inevitably confronted with the question of how to reduce the risk of a second stroke. In addition to the risk of recurrent stroke, a stroke survivor is also at risk of suffering acute myocardial infarction (MI) and other cardiovascular complications. Efforts to reduce cardiovascular risk may potentially also reduce stroke risk.

Physical activity as contrasted to sedentary lifestyle is associated with a reduced risk of first stroke, but in one of these studies the reduction in stroke risk did not reach statistical significance. In a Norwegian study the relative risk of stroke mortality was 0.56 (95% confidence interval [CI] 0.36 - 0.88) in physically active women aged 70-79 years, compared to women with lower physical activity.

Purpose of the ExStroke Trial:

To evaluate the effect of instruction in physical training on "Physical Activity Scale for Elderly" (PASE)in patients with ischemic stroke.

Other endpoints are recurrent stroke, MI, death of all causes, and vascular death after an ischaemic stroke in patients randomised to receive verbal instruction by a stroke physician/a neurologist and a physiotherapist concurrently with written information on physical exercise versus a control group, which is to receive standard information on the usefulness of physical activity. Both groups will receive physiotherapy according to the usual standards of the department to which the patients are admitted.

The Interventions:

Physical exercise after discharge from hospital:

Patients randomised to the physical exercise group shall have a session with a stroke physician/a neurologist, and a physiotherapist in which the patient's possibilities and wishes of training activity after discharge are discussed. In agreement with the patient, a training program is designed for the individual patient according to the patient's resources and capability. The training program on which the patient, the physician, and the physiotherapist have agreed must be written down; the patient will keep a copy of the training program, another copy is kept in the patient files, and a third copy is kept in Clinical Record Form (CRF).

At the follow-up visits the level of physical activity is evaluated using the "Physical Activity Scale in the Elderly" (PASE) in both groups and the Copenhagen City Heart Study questionnaire on physical activity.

It is recommended that patients in the active group should be contacted between the follow-up sessions by the physiotherapist in order to stimulate physical exercise. Patients in the control group shall receive the same high quality medical care, but without further discussion of physical training, unless the patient requests such information.

Hypotheses:

Several studies have shown that a certain amount of physical activity is associated with reduced risk of first-ever stroke. It is hypothesised that a certain level of physical exercise in patients with ischaemic stroke, will reduce the risk of subsequent cardio-vascular events. The following hypotheses will be tested:

* Level of physical activity will increase when patients are instructed in a physical training program.
* The incidence of recurrent stroke, MI, or death following an ischaemic stroke will be lower in patients who have received verbal and written instruction on physical exercise compared with those in the control group.

Outcome Measures

Primary Outcome Measure: physical activity as measured by PASE

Secondary Outcome Measure: time from randomisation to recurrent stroke, or to MI, or to death of all causes.

Third Outcome Measure: time from randomisation to recurrent stroke, MI and vascular death.

Fourth Outcome Measure: frequency of recurrent stroke.

Fifth Outcome Measure: activities of daily living as measured by modified Rankin Scale.

Sixth Outcome Measure: quality of life

Seventh Outcome Measure: frequency of falls and fractures.

Study Design:

Consecutive patients, meeting all inclusion criteria, and none of the exclusion criteria, will be asked if they want to participate in the trial. Patients will be included as soon as convenient and within 90 days after onset of an ischaemic stroke. There will be follow-up sessions at 3,6, 9, 12, 18, 24 months. The study is a randomised, single blind, parallel group, multicenter, international clinical trial.

Informed Consent:

Randomisation:

The randomisation will be performed centrally with randomisation in blocks 1:1, stratifying for center, sex, age, and stroke severity. The Copenhagen Trial Unit (CTU) will perform the randomisation.

Study Population and Planned Sample Size:

Patients with ischaemic stroke being 40 years of age or older will be included in the study. It is unknown, if level of physical activity can be increased by repeated information given to patients with a stroke. Level of physical activity is evaluated according to the PASE scale, which is expected to be approximately 70 as a mean value. Based on a standard deviation of 50, a minimal relevant difference of 20 in PASE score, a Type I error of 5%, a Type 2 error of 20%, it is estimated that 100 patients should be included in each of the two study arms. To take into account withdrawals and dropouts, about 50% more patients should be included in each arm, giving a total of 300 patients in the pilot trial.

Inclusion Criteria:

* Subjects aged 40 years or older.
* Patients with a clinical diagnosis of stroke; symptoms lasting 24 hours or more.
* CT-scan of the brain must either show a new infarct or be normal. Patients only with infarcts without clinical symptoms cannot be included.
* Inclusion shall take place before day 90 after stroke onset.
* Informed consent after verbal and written information.
* The patient must be able to walk either unaided or with a cane or a walker.

Exclusion Criteria:

* Patients who are unable to understand the information, or who can not cooperate, are excluded.
* Patients confined to a wheelchair or bed.
* CT-scanning showing intracranial haemorrhage or focal pathology other than infarction, cerebral atrophy, or leucoaraiosis.
* Modified Rankin score of 4 or 5 before the actual stroke.
* Serious medical disease such as AIDS, metastatic cancer, or abnormalities that the investigator feels may compromise the patient's successful participation in the trial.
* Earlier randomisation in this trial.

Baseline Registration:

* Sex and birthday
* Date of qualifying stroke (day, month, year)
* Type of stroke
* Results of CT scan, ECG, and Doppler examination of carotid arteries shall be obtained
* Information on treatment with anti-thrombotic medication and on treatment with anti-hypertensive medication before discharge of the index stroke
* Information on blood pressure on inclusion
* Weight and height

Adverse Events:

Stroke patients are at risk of adverse events such as the occurrence of falls, fractures.

Follow-Up Visits:

Follow-up examinations take place at 3, 6, 9, 12, 18 and 24 months after the inclusion of the patient in the trial. On each visit the medical history shall include information on date of recurrent stroke, date of transient ischaemic attacks (TIA), date of gastro-intestinal bleeding, other bleeding episodes, and date of MI, falls, and fractures, and date of any serious adverse events.

In case of hospital admissions, information on diagnosis and length of stay shall be obtained.

In case of death, information on date of death shall be retrieved and the cause of death be given as either baseline stroke, new stroke, cardiac disease, vascular causes, or other causes.

On each follow-up visit the patients randomised to "physical exercise group" shall have repeated instruction by the physiotherapist as to the exercises suggested at baseline, or adapted to the present capability of the patient. Such adapted instructions on the training program must be written down. The patient shall receive a copy of it, a second copy shall be inserted in the patient record, and a third copy in the case record form.

On each visit in all patients the physical activity scale (PASE) shall be completed. The interview will be done by a co-investigator, who is blinded as to what group the patient was randomised.

Three Month Follow-Up:

Information is recorded on the following items:

* Scandinavian Stroke Scale
* Modified Rankin Scale
* Blood pressure
* Tobacco smoking
* Alcohol consumption
* Antithrombotic medication
* Antihypertensive medication
* PASE form
* Events such as recurrent stroke, MI, or adverse events are recorded
* Quality of life form

  6, 9, 12, 18 and 24 Month Follow-Ups: Information is recorded as three months follow-up.

Ethical Considerations:

It is unknown whether physical exercise will influence the rate of recurrent vascular events, MI, and mortality after an ischaemic stroke. It is, however, assumed that physical activity may favourably influence the prognosis. Therefore, all patients in the trial will be advised as to a healthy lifestyle including the possible benefit of physical exercise. Those, who are randomised to the active group, will in addition receive special instruction by the physiotherapist and a physician. The trial shall be accepted by the local ethics committees and informed, written consent is a requirement for participation in the study. Participation is voluntary and the patients can choose to withdraw from the study at any time.

Outcome Event Adjudication Committee:

The outcome event adjudication committee will blindly evaluate and adjudicate events such as death, causes of death, recurrent stroke, MI and traumatic event or other adverse events.

The Independent Data Safety and Monitoring Board (DSMB):

DSMB will receive blinded data from the Trial Data Center. The DSMB will evaluate events such as death, causes of death, recurrent stroke, MI, and adverse effects. The DSMB may advise early interruption of the trial if analyses demonstrate significant difference in the occurrence of secondary outcome measures with p < 0.001 between group A and group B.

The DSMB will also follow the development of serious adverse events occurring in the 2 intervention arms of the trial.

Finance and Insurance:

Financial support for the study will be applied for in national private and public funds. Insurance will follow national regulations.

Publication Policy:

The main publication will be submitted to a major peer reviewed international journal. All investigators, who are not included as co-authors, will be acknowledged in an appendix.

ELIGIBILITY:
Inclusion Criteria:

* Subjects aged 40 years or older.
* Patients with a clinical diagnosis of stroke; symptoms lasting 24 hours or more.
* Computed tomography (CT)-scan of the brain must either show a new infarct or be normal. Patients only with infarcts without clinical symptoms cannot be included.
* Inclusion shall take place before day 90 after stroke onset.
* Informed consent after verbal and written information.
* The patient must be able to walk either unaided or with a cane or a walker.

Exclusion Criteria:

* Patients who are unable to understand the information, or who cannot cooperate, are excluded.
* Patients confined to a wheelchair or bed.
* CT-scanning showing intracranial haemorrhage or focal pathology other than infarction, cerebral atrophy, or leucoaraiosis.
* Modified Rankin score of 4 or 5 before the actual stroke.
* Serious medical disease such as AIDS, metastatic cancer, or abnormalities that the investigator feels may compromise the patient's successful participation in the trial.
* Earlier randomisation in this trial.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 314 (Actual)
Dates: Start 2003-09; Study Completion 2007-10 (Actual)

PRIMARY OUTCOMES:
Difference in physical activity scale for the elderly | 24 months

SECONDARY OUTCOMES:
Occurrence of stroke, MI or death | 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Gudrun Boysen, MD, Principal Investigator — Dept. of Neurology, Bispebjerg Hospital
Locations (1):
- Bispebjerg Hospital, Copenhagen, Denmark

REFERENCES:
- [Derived] Boysen G, Krarup LH, Zeng X, Oskedra A, Korv J, Andersen G, Gluud C, Pedersen A, Lindahl M, Hansen L, Winkel P, Truelsen T; ExStroke Pilot Trial Group. ExStroke Pilot Trial of the effect of repeated instructions to improve physical activity after ischaemic stroke: a multinational randomised controlled clinical trial. BMJ. 2009 Jul 22;339:b2810. doi: 10.1136/bmj.b2810. PMID 19900934
- [Derived] Krarup LH, Gluud C, Truelsen T, Pedersen A, Lindahl M, Hansen L, Michelsen S, Andersen G, Zeng X, Korv J, Oskedra A, Boysen G; ExStroke Pilot Trial Group. The ExStroke Pilot Trial: rationale, design, and baseline data of a randomized multicenter trial comparing physical training versus usual care after an ischemic stroke. Contemp Clin Trials. 2008 May;29(3):410-7. doi: 10.1016/j.cct.2007.09.008. Epub 2007 Oct 9. PMID 18029233